CLINICAL TRIAL: NCT03613402
Title: BRAVO - Betrixaban Registry Using Real Time Observations in Acute Medical Illness to Assess Venous Thrombosis and Bleeding Outcomes
Status: Withdrawn | Type: Observational
Why Stopped: Due to slow enrollment.
Sponsor: Portola Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Other Study IDs: 18-025
Record Dates: First submitted 2018-07-19; First posted 2018-08-03 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Venous Thromboses
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Patients at risk of VTE who are prescribed betrixaban to prevent VTE
- Cohort 2: Patients at risk of VTE who are prescribed betrixaban or other VTE prophylaxis

SUMMARY:
Part 1 - Evaluate the real-world implementation of extended prophylaxis with betrixaban in the acutely ill hospitalized medical population Part 2 - Describe patterns of Venous thromboembolism (VTE) prophylaxis in acutely ill medical patients who qualify for extended VTE prophylaxis

ELIGIBILITY:
Inclusion Criteria:

-Part 1 -

1. Hospitalized acutely ill medical patient
2. Patient prescribed betrixaban
3. Signed informed consent

Part 2 -

1. Hospitalized acutely ill medical patient
2. Patient prescribed betrixaban OR must satisfy criteria a and b:

   1. Moderately or severely restricted immobility: patient restricted to bed for at least 24 hours (severe) or restricted to bed for at least 12 hours (moderate) during their hospitalization
   2. At least One additional risk factor:

Age > 70 years D-dimer > 2x institutional Upper Limit of Normal (ULN) Obesity: Body mass index (BMI) > 30 kg/m2) History of pulmonary embolism (PE) or deep venous thrombosis (DVT) Active cancer (diagnosed, treated, or progressing in the past 6 months) History of thrombophilia Recent trauma or surgery (within 30 days prior to admission) Ongoing hormonal treatment ICU stay 3. Signed informed consent

Exclusion Criteria:

* Part 1 - 1. High bleeding risk - any of the following:

  1. Patient on dialysis
  2. Low platelet count (<50 per 109/L)
  3. Known bleeding disorder (congenital or acquired)
  4. Liver disease prohibitive to anticoagulation
  5. Bleeding within last 30 days
  6. Use of Dual Anti-Platelet Therapy (DAPT)

Part 2

1. Patients who are on another oral anticoagulant (OAC) for any reason at the time of hospitalization and will remain on it
2. Condition requiring use of OAC at admission, other than VTE prophylaxis (eg, acute VTE at admission)
3. High bleeding risk any of the following:

   1. Patient on dialysis
   2. Low platelet count (<50 per 109/L)
   3. Known bleeding disorder (congenital or acquired)
   4. Liver disease prohibitive to anticoagulation
   5. Bleeding within last 30 days
   6. Use of Dual Anti-Platelet Therapy (DAPT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acutely ill medical patients, hospitalized, prescribed therapy for VTE prophylaxis and who would qualify for extended prophylaxis (whether or not they receive prophylaxis).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Thrombotic Events at 45 days: VTE, MI, Stroke, Transient ischemic attack (TIA) | 45 days
  Thrombotic Events at 45 days: VTE, MI, Stroke, TIA

SECONDARY OUTCOMES:
Bleeding rates at 45 days | 45 days
  Bleeding rates at 45 days

CONTACTS AND LOCATIONS:
Locations (1):
- Durham, Durham, North Carolina, United States